CLINICAL TRIAL: NCT03152721
Title: Interventional Study of the Effect of Parkinson Kinetigraph Recordings on the Clinical Management and Outcome in Parkinson's Disease
Brief Title: The Effect of Parkinson Kinetigraph Recordings on the Management and Outcome in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Filip Bergquist, Associate Professor, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WestPORTSintervention; PARKreg (Registry Identifier: Svenska Parkinsonregistret)
Record Dates: First submitted 2017-05-10; First posted 2017-05-15 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Parkinson Disease
Keywords: accelerometry; home based; motor complications; Parkinson KinetiGraph; Registry
MeSH Terms: conditions — Parkinson Disease | interventions — Diagnostic Self Evaluation

STUDY DESIGN:
Intervention Model Description: 1:1 randomisation to intervention and control group. The effect of providing the objective measurement and self assessment scales compared to only self assessment scales on the management decisions will be evaluated. A secondary outcome is the ability of the measurement to identify sub-optimally treated individuals in comparison with self assessment scales.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patient not aware of which information has been provided to his/her physician. Post data collection the groups will be assigned coded group names so that the conditions are masked to the assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Placebo Comparator): Treating physician will in advance of upcoming visit be provided with the self assessment scales PDQ8 and NMS-Questionnaire to aid clinical assessment
  Interventions: Other: Self assessment
- Intervention (Experimental): Treating physician will in advance of upcoming visit be provided with a Parkinson KinetiGraph recording report and interpretation in addition to the self assessment scales PDQ8 and NMS-Questionnaire to aid clinical assessment
  Interventions: Device: Parkinson KinetiGraph; Other: Self assessment

INTERVENTIONS:
Device: Parkinson KinetiGraph — The Parkinson Kinetigraph (PKG) is a wrist-worn accelerometer shaped as a watch. It records spontaneous movements and for every two minutes provides a bradykinesia score and a dyskinesia score. Furthermore it analysis movement for tremor-like episodes and registers the time with tremulous movements as well as time with extreme immobility suggesting sleep. The device can be programmed with drug intake times and provide a reminder signal. Intake of drug can be indicated on the device.
  Other Names: Parkinson KinetiGraph Mk II; PKG
  Arms: Intervention
Other: Self assessment — Administration of self assessment questionnaires are made within 2 weeks from starting a PKG recording. The assessments are Parkinson Disease Quality of life 8 question short version and the Non Motor Symptom in Parkinson Disease Questionnaire.
  Other Names: PDQ8; NMS-Questionnaire

SUMMARY:
With time most people with Parkinson's disease (PwP) develop fluctuations in motor symptoms in relation to medication intake. The prevalence may be both under and overestimated as it is based on history rather than observation. Patterns in fluctuations are difficult to determine and it has been demonstrated that every 30-minute diaries need to be kept for 10 days or more to safely represent fluctuation patterns. The Parkinson Kinetigraph (PKG) is an automated system that is carried passively and provides similar information after wearing the device for 6 days. Clinical experience is that most patients agree that results are representative to their experiences. It is not known if using the PKG routinely at any stage of PD will change management of the disease. The hypothesis of this study is that providing PKG information to neurologists will lead to a more active management that may improve outcome in PD patients.

DETAILED DESCRIPTION:
Patients that have previously not performed a PKG recording will be recruited from the WestPORTS community based cohort of outpatients with PD in West Sweden. The WestPORTS study includes self-assessments like PDQ8 and NMS-Q as well as PKG recordings. On inclusion in WestPORTS-Int subjects will be randomized by minimization for age, gender and disease duration into one of two study arms. In the intervention group the PKG recording of the subject will be made available, together with a summarized interpretation, to the subject's regular neurologist/geriatrician before the next scheduled visit/contact. The neurologist will also be provided with PDQ8 and NMS-Q responses. In the control group only PDQ8 and NMS-Q responses will be available to the treating neurologist/geriatrician.

At the next regular visit/contact the physician will fill out an assessment of the state of the patient, whether stable or in need of change in management. Any contraindications to changed management will be noted and the decision to change or not change management will be recorded as the primary outcome of the study. Secondary outcomes are the patient reported experience of outpatient care according to a modified version of the Generic Short Patient Experiences Questionnaire (GS-PEQ), as well as patient reported (PDQ8, NMS-Q, PRO-PD, EQ5D5L) and PKG outcomes at a time point three months later.

Change of management is defined as any of the following:

1. Adding or stopping a dopamine agonist, COMT- or MAO-inhibitor, anticholinergic or amantadine.
2. Fractionation or de-fractionation of the current daily levodopa dose
3. Change of current Levodopa Equivalent daily dose by 15% or more
4. Start or stop of night medication
5. Referral for device assisted therapy (LCIG, apomorphine pump or DBS)

Actual change of management (as opposed to decision to change) will be documented by retrospective review of medical records and prescription records. This will be a secondary measure.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of Parkinson's disease (ICD G209) according to medical records
2. A visit to an outpatient neurological or geriatric clinic in the region Vastra Gotaland, Sweden within the last -1 to -7 months according to medical records.
3. Randomized to invitation to participate in the WestPORTS objective measurement Cohort study (NCT03130595) by 1:4 randomization based on the full population fulfilling criteria 1 and 2.
4. Written informed consent
5. No previous PKG recording has been performed with the subject.

Exclusion Criteria:

1. Withdrawal of consent.
2. Unable to wear a PKG on either wrist.
3. The patient's physician is the PI of the study (F Bergquist)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2017-04-30 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Decision to change management | On first regular contact, RC, (telephone or visit) wich takes place within four months after PKG-recording
  The decision to change management of Parkinson's disease as reported by the treating physician.
  Change of management is defined as any of the following:
  1. Adding or stopping a dopamine agonist, COMT- or MAO-inhibitor, anticholinergic or amantadine.
  2. Fractionation or de-fractionation of the current daily levodopa dose
  3. Change of current Levodopa Equivalent daily dose by 15% or more
  4. Start or stop of night medication
  5. Referral for device assisted therapy (LCIG, apomorphine pump or DBS)

SECONDARY OUTCOMES:
Actual change of management | Change should take place within 4 weeks from the RC.
  A retrospectively verified (medical and prescription records) change in management of PD as defined in the primary variable
Patient Reported Experience of Care | The assessment will be made within 3 days from the first RC after PKG-recording,
  A modified version of Generic Short Patient Experiences Questionnaire (GS-PEQ), Sjetne et al 2011 will be used. The modified questionnaire has 13 questions that are answered with a 5 grade Likert scale and a 5 grade Likert scale describing the importance of each question. Items will be analyzed separately as well as as summary scores
PRO-PD score at 3 months after the first regular visit | The assessment is made 3 months after the RC.
  The Patient Reported Outcome in PD web questionnaire will be reported as summary score as well as per symptom domain.
PDQ-8 score at 3 months after the first regular visit | The assessment is made 3 months after the RC.
  The 8 question version of Parkinson Disease Quality of Life Questionnaire. Reported as index score (0-100%)
NMSQ score at 3 months after the first regular visit | The assessment is made 3 months after the RC.
  The Non Motor Symptoms Questionnaire will be administered and the number of reported symptoms within the last month are reported
EQ5D-5L at 3 months after the first regular visit | The assessment is made 3 months after the RC.
  The EuroQoL 5 dimension 5 level scale of generic health
Parkinson Kinetigraph bradykinesia measurement at 3 months after the first regular visit | The assessment is made 3 months after the RC.
  Median BK score of a 6 day recording.
Parkinson Kinetigraph dyskinesia measurement at 3 months after the first regular visit | The assessment is made 3 months after the RC.
  Median DK score of a 6 day recording.
Parkinson Kinetigraph fluctuation score at 3 months after the first regular visit | The assessment is made 3 months after the RC.
  Fluctuation dyskinesia score (FDS) of a 6 day recording.
Parkinson Kinetigraph Tremor measurement at 3 months after the first regular visit | The assessment is made 3 months after the RC.
  Mean percent day-time (9-18) tremor time in a 6 day recording.
Parkinson Kinetigraph immobility measurement at 3 months after the first regular visit | The assessment is made 3 months after the RC.
  Mean percent day-time (9-18) immobility time in a 6 day recording.
Change in PDQ8 compared to baseline | Assessed 3 months after the RC and at end of study 12 months after inclusion visit
  The change in PDQ8 index score compared to the baseline assessment that is made at the inclusion visit
Change in NMSQ compared to baseline | Assessed 3 months after the RC and at end of study 12 months after inclusion visit
  The change in number of reported non-motor symptoms characterized as improvement, no change, or deterioration compared to the baseline assessment that is made at the inclusion visit
Change in EQ5D5L compared to baseline | Assessed 3 months after the RC and at end of study 12 months after inclusion visit
  The change in index score characterized as improvement, no change, or deterioration compared to the baseline assessment that is made at the inclusion visit
Change in Parkinson Kinetigraph bradykinesia score compared to baseline | Assessed 3 months after the RC and at end of study 12 months after inclusion visit
  The change in BK score characterized as improvement, no change, or deterioration compared to the baseline assessment that is made at the inclusion visit. Improvement defined as abnormal score that has changed to within normal limits, no change defined as normal score that remains within normal limits and deterioration defined as normal score that changes to a score outside normal limits
Change in Parkinson Kinetigraph dyskinesia score compared to baseline | Assessed 3 months after the RC and at end of study 12 months after inclusion visit
  The change in DK score characterized as improvement, no change, or deterioration compared to the baseline assessment that is made at the inclusion visit. Improvement defined as abnormal score that has changed to within normal limits, no change defined as normal score that remains within normal limits and deterioration defined as normal score that changes to a score outside normal limits
Change in Parkinson Kinetigraph fluctuation score compared to baseline | Assessed 3 months after the RC and at end of study 12 months after inclusion visit
  The change in FDS score characterized as improvement, no change, or deterioration compared to the baseline assessment that is made at the inclusion visit. Improvement defined as abnormal score that has changed to within normal limits, no change defined as normal score that remains within normal limits and deterioration defined as normal score that changes to a score outside normal limits
Change in Parkinson Kinetigraph Tremor measurement compared to baseline | Assessed 3 months after the RC and at end of study 12 months after inclusion visit
  The change in percent tremor time characterized as improvement, no change, or deterioration compared to the baseline assessment that is made at the inclusion visit. Improvement defined as a decrease in tremor time which was higher than 0.9% at baseline, no change defined as tremor time that remains lower or equal to 0.9% or remains the same as at baseline. Deterioration defined as an increase in tremor time that results in a tremor time higher than 0.9% at follow up.
Change in Parkinson Kinetigraph Immobility measurement compared to baseline | Assessed 3 months after the RC and at end of study 12 months after inclusion visit
  The change in percent immobility time characterized as improvement, no change, or deterioration compared to the baseline assessment that is made at the inclusion visit. Improvement is defined as a decrease in immobility time, no change is defined as immobility time that remains the same as at baseline. Deterioration defined as an increase in immobility time at follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Filip Bergquist, Principal Investigator — Göteborg University
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided